CLINICAL TRIAL: NCT06208007
Title: Arterial Stiffening as a Predictor for Diastolic Cardiac Dysfunction and HFpEF
Acronym: ARTSPREDICTION
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Alexander Schulz, Principal Investigator, University Medical Center Goettingen
Other Study IDs: 9/12/23
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Cardiovascular Morbidity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood samples, urine samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients at risk for developing heart failure with preserved ejection fraction (HFpEF) will undergo a structured clinical assessment, transthoracic echocardiography and pulse-wave analysis to investigate the association of arterial stiffening and the development of cardiac diastolic dysfuntion and HFpEF.

ELIGIBILITY:
Inclusion Criteria:

One or more of the following criteria:

* Age > 60 years
* Arterial hypertension (RR systolic ≥ 140 mmHg or diastolic ≥ 90 mmHg or ≥ 2 antihypertensive drugs)
* Diabetes mellitus Type I or II
* Atrial fibrillation
* Chronic kidney disease (GFR < 60 ml/min/1,73 m2 or urine albumin ≥ 30mg/24h or ACR ≥ 30 mg/g)
* BMI ≥ 30 kg/m2
* NYHA ≥ II
* E/e' > 8

Exclusion Criteria:

* Left ventricular ejection fraction < 50 %
* Significant valve disease (Grade III or higher)
* History of interventional or surgical valve repair
* Regional wall motion abnormalities
* Respiratory diseases as a known cause for dyspnea
* Atrial flutter or fibrillation during examination
* Hypertrophic/restrictive/arrhythmogenic/dilatative cardiomyopathies including cardiac amyloidosis or sarcoidosis and toxic cardiomyopathy
* History of heart transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients at risk for HFpEF
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in HFA-PEFF-Score | 24 months
  Heart Failure Association - Pre-test assessment, Echocardiography and Natriuretic Peptide, Functional testing, Final aetiology; 2-4 points: Diastolic Stress Test or Invasive Haemodynamic Measurements recommended; ≥ 5 points: HFpEF [min. 0 points, max. 6 points]
Development of HFpEF | 24 months
  Defined as ≥ 5 points in HFA-PEFF-Score Heart Failure Association - Pre-test assessment, Echocardiography and Natriuretic Peptide, Functional testing, Final aetiology; 2-4 points: Diastolic Stress Test or Invasive Haemodynamic Measurements recommended; ≥ 5 points: HFpEF [min. 0 points, max. 6 points]
Composite endpoint cardiovascular events | 24 months
  Cardiovascular hospitalisation or death

SECONDARY OUTCOMES:
Change of individual parameters included in the HFA-PEFF-Score | 24 months
  Heart Failure Association - Pre-test assessment, Echocardiography and Natriuretic Peptide, Functional testing, Final aetiology; 2-4 points: Diastolic Stress Test or Invasive Haemodynamic Measurements recommended; ≥ 5 points: HFpEF [min. 0 points, max. 6 points]
Change of NT-proBNP | 24 months
Change of NYHA-class | 24 months
Development or aggravation of albuminuria | 24 months
Change of blood-creatinine | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsmedizin Göttingen, Göttingen, Lower Saxony, Germany